CLINICAL TRIAL: NCT03075943
Title: Efficacy of a Brown Seaweed Extract on Glycemic Control and Body Weight in Overweight Pre-diabetic Subjects.
Brief Title: Brown Seaweed Extract on Glycemic Control and Body Weight
Acronym: Algues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Ministry of Agriculture, Fisheries and Food, Quebec (Other Government); innoVactiv Inc. (Industry)
Responsible Party: Principal Investigator, Helene Jacques, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ALGUES 2016-227
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: PreDiabetes; Insulin Resistance
MeSH Terms: conditions — Prediabetic State; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- InSea2 (Experimental): 2 capsules/day of InSea2 administered 30 min before a meal (breakfast, lunch or diner) combined with weight loss program (individualized nutritional intervention with a daily restriction of 500 kcal)
  Interventions: Dietary Supplement: InSea2
- Placebo (Placebo Comparator): 2 capsules/day of Placebo administered 30 min before a meal (breakfast, lunch or diner) combined with weight loss program (individualized nutritional intervention with a daily restriction of 500 kcal)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: InSea2 — Daily supplement: 2 capsules of InSea2
  Other Names: Brown seaweed extract supplement
  Arms: InSea2
Dietary Supplement: Placebo — Daily supplement: 2 capsules of Placebo
  Other Names: Control
  Arms: Placebo

SUMMARY:
The overall goal of this study is to investigate the effects of a daily dietary supplement of brown seaweed (2 capsules of InSea2®) on body weight, glycemic control and insulin secretion in overweight prediabetic men and women in association with a moderate weight loss intervention.

DETAILED DESCRIPTION:
Diets that produce lower glucose and insulin responses may reduce diabetes and cardiovascular risk. They may also facilitate weight control by promoting satiety, insulin sensitivity and optimal insulin secretion after a meal. Food ingredients may indeed reduce postprandial glucose and insulin response through an inhibition of α-amylase and α-glucosidase activity that may slow down the absorption of carbohydrates. InSea2® is a unique combination of polyphenolic extracts of brown algae (Ascophyllum nodosum and Fucus vesiculosus) which has been shown to inhibit the action of α-amylase and α-glucosidase. Preliminary data in healthy men and women have demonstrated a reducing effect on plasma insulin of a single intake of InSea2® consumed with a high-carbohydrate meal.

The main objective is to evaluate the effects of a daily dietary supplement of 500 mg (2 capsules) of brown algae extract powder (InSea2®) on body weight and blood glucose homeostasis (glucose, insulin, c-peptide) measured in the fasting state and during a 2-hour oral glucose tolerance test (OGTT) in overweight prediabetic men and women.

The secondary objectives are to assess the contribution of a daily consumption of this supplement (InSea2®) on weight loss when associated with a daily caloric restriction of 500 kcal due to individualized nutritional intervention on markers of lipid profile, blood pressure, inflammation, oxidative stress and gut barrier integrity.

The investigators expect that InSea2® lowers body weight and blood glucose homeostasis (glucose, insulin or C-peptide, as marker of insulin secretion, in the fasting state or during a 2-hour oral glucose tolerance test) in association with metabolic and inflammatory markers in the context of moderate weight loss in overweight prediabetic human subjects.

ELIGIBILITY:
Inclusion Criteria:

* overweight (BMI > 25; waist circumference ≥ 80cm for women and ≥ 94 cm for men)
* fasting insulin (≥ 60 pmol/L)
* Impaired fasting glycemia with or without impaired glucose tolerance
* HbA1c between 5.6 and 6.4
* non-smoking
* stable weight in the past 3 months

Exclusion Criteria:

* diabetes
* chronic disease (thyroid dysfunction, hepatic or gastrointestinal disorder, uncontrolled hypertension)
* taking drugs that could affect glucose or lipid metabolism or weight and appetite
* taking dietary supplements (protein powders, fish oil, omega-3 or any marine supplements) or natural health products that could affect glucose, lipid, weight or appetite
* major surgery 3 months prior to the study
* pregnancy
* fish, seafood or iodine allergy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in blood glucose (mmol/L) | at baseline and at the end of the intervention (12 week)
  glucose in the fasting state and during a 2h-OGTT
Changes in blood insulin (pmol/L) and C-peptide (pmol/L) | at baseline and at the end of the intervention (12 week)
  insulin and C-peptide in the fasting state and during a 2h-OGTT
Changes in anthropometrics | at baseline and at the end of the intervention (12 week)
  body weight (kg), lean mass (kg) and fat mass (kg)

SECONDARY OUTCOMES:
Changes in blood pressure | at baseline and at the end of the intervention (12 week)
  Systolic and diastolic blood pressure (mmHg)
Changes in heart rate | at baseline and at the end of the intervention (12 week)
  Heart rate (n/min)
Changes in lipid profile | at baseline and at the end of the intervention (12 week)
  cholesterol (mmol/L), triglycerides (mmol/L), LDLc (mmol/L), HDLc (mmol/L)
Changes in hsCRP | at baseline and at the end of the intervention (12 week)
  HsCRP (mg/L)
Changes in Il-6 | at baseline and at the end of the intervention (12 week)
  IL-6 (pg/L)
Changes in marker of oxidative stress | at baseline and at the end of the intervention (12 week)
  F2-isoprostane (ng/mL)
Changes in markers of gut barrier integrity | at baseline and at the end of the intervention (12 week)
  LBP (ng/mL), zonulin (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Jacques, PhD, Principal Investigator — Institue of Nutrition and Functional Food (INAF), Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Laval University, Québec, Canada